CLINICAL TRIAL: NCT05314894
Title: The Effect of the Program Based on the PRECED-PROCEED Model "I am Giving up Smoking, I am Protecting My Future and My Health" on Smoking Behaviour of Nursing Students
Brief Title: The Effect of the Education Program Based on the PRECEDE-PROCEED Model on the Smoking Behaviors of Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Erdal Akdeniz, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AhiEvranU_EAkdeniz_001
Record Dates: First submitted 2022-01-01; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Smoking Cessation
Keywords: Nursing Students; Stopping Smoking
MeSH Terms: conditions — Smoking Cessation | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- initiative group (Experimental): The first session will be right after the pre-test, the second session will be 15 days after the first session, and the last session will be 15 days after the second session. After the training is over, a total of 40 messages will be sent to the students in the initiative group, taking into account the factors that affect, strengthen and activate the main communication via the WhatsApp program.
  Interventions: Behavioral: Education
- control group (No Intervention): No intervention will be made

INTERVENTIONS:
Behavioral: Education — Giving training to the students in the initiative group to quit smoking in three sessions, sending messages via whatsapp program and telephone counseling
  Arms: initiative group

SUMMARY:
The causes of death due to smoking are responsible for 11.5% of the total deaths in the world. Smoking causes lung cancer, chronic obstructive pulmonary disease (COPD), ischemic heart disease and cerebrovascular diseases. In some studies on nursing students in the world, the prevalence of smoking is between 13.9% and 32%; It is known that it varies between 12.9% and 28% in Turkey. At the end of this study, nursing students are supported in smoking cessation by providing smoking cessation training, they become a role model for the society by gaining the right behavior, creating a society that smokes less, reducing the financial burden on the state as a result of protecting individuals from possible chronic diseases, and guiding health trainings on this subject. It is foreseen that it will be a guide in its implementation in the whole country. The aim of this study is to determine the effect of the I Stop Smoking, Protecting My Future and Health program based on the Preced-Proceed Model on the smoking behavior of nursing students.

DETAILED DESCRIPTION:
This study will be conducted in non-randomized groups in a quasi-experimental fashion as pre-test-post-test.

The population of the research was formed by the students in the Nursing Department of the Faculty of Health Sciences of Kırşehir Ahi Evran University. There are two branches of daytime education and two branches of secondary education, and the total number of students in the nursing department is 802. The sample size of the study was calculated using the G*Power (v3.1.9.6) package program. The power of the study was 80% and the sample size was α =0.05; It was calculated as a total of 64 people, 32 of which were interventions and 32 were control groups. However, considering the losses, 20% more than the calculated value was included in the sample and it was planned to include a total of 80 students, 40 of whom were in the intervention group and 40 in the control group.

Selection and Assignment of Individuals to the Intervention and Control Group Before being divided into intervention and control groups, students' consent was obtained and a pre-test was applied. Formal education and secondary education students were coded as A and B. For example, formal education A, secondary education B. The students in the related group were stratified by gender and the layer weight was determined. Random numbers were created in the Excel program and it was determined who would be in the groups with the simple random sampling method. In addition, which of the previously coded groups A and B would be the intervention group and which one would be the control group was determined by drawing lots. All these procedures were carried out by a person other than the researcher. Thus, it was determined who would be in the intervention and control group, and it was explained to the researcher before the training whether group A or group B was the intervention or control group.

Dependent variables:

* Behavior modification level
* Decision equilibrium level
* Self-efficacy level
* Level of encouraging factors
* Level of stages of change
* Number of people who quit smoking
* Nicotine addiction level
* Health perception level

Independent variables:

"I Stop Smoking, I Protect My Future and My Health" program based on the PRECEDE-PROCEED Model.

As data collection tools; Smoker identification form, individual information form, Behavior change process scale, Decision balance scale, Self-efficacy scale, Encouraging factors scale, Classification of stages of change scale, Fagerström nicotine addiction test will be used. The data were also planned to be collected in this environment before the first training (pretest), and after the second and third training (posttest). The first session will be held immediately after the pre-test, the second session will be held 15 days after the first session, and the last session will be held 15 days after the second session. A total of 40 messages will be sent to the students in the initiative group through the WhatsApp program, taking into account the factors that affect, strengthen and enable the main

ELIGIBILITY:
Inclusion Criteria:

* Approving to participate in the study,
* Smoker (according to WHO, a person who smokes at least one cigarette per day),
* According to the Fagerström Test for Nicotine Dependence, nicotine addiction is at least "very low" or higher*,
* Not having any communication barriers to participate in the study,
* Those who are in the stages of "thinking" and "preparation" of the stages of change according to the Classification of Stages of Change Scale for smoking cessation**,
* Not taking any smoking cessation treatment at the time of the study,
* Having a smart mobile phone and using the WhatsApp program,
* Consists of students who have not received training in smoking cessation before

Exclusion Criteria:

* Non-smokers
* Those who do not plan to quit smoking (those who are at the stage of "not thinking" according to the Classification of Stages of Change Scale)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
It is expected that the students in the intervention group will be more likely to quit smoking than the students in the control group. | 6 months
  Determining the number of non-smokers, unit of measure: frequency, scale of stages of change, Individual information form
The level of nicotine addiction in the intervention group is expected to be lower than in the control group. | 6 months
  Measuring nicotine addiction, unit of measure: nicotine addiction level, Fagerström Test for Nicotine Dependence

SECONDARY OUTCOMES:
The level of behavior change is expected to be higher in the intervention group than in the control group. | 6 months
  Measuring behavior change, comparison of scale tools between groups. Name of the scale: Behavior Change Processes Scale. A maximum of 110 and a minimum of 22 points are obtained from the scale. A high score on this scale is interpreted as a high chance of success in behavior change, and a low score is interpreted as a low chance of success.
It is expected that there will be a higher level of decision balance in the intervention group than in the control group. | 6 months
  Measurement decision balance, Comparison of scale averages between groups. Name of the scale: Decision Balance Scale. The scale consists of 12 questions about the negative aspects of smoking and 12 questions about the positive aspects of smoking. The total score of the scale is calculated by subtracting the perceived harm total score from the perceived benefit total score of smoking, and a negative (-) result indicates that the perceived harms of smoking dominate in the decision balance and a positive (+) result. shows that the perceived benefits of smoking are more in the decision balance. A minimum of 12 and a maximum of 60 points can be obtained for both sub-dimensions. A high score on the questions about the positive aspects of smoking indicates that he is undecided in changing behavior, and a high score on the negative aspects indicates that he is determined to change and maintain the behavior.
Higher self-efficacy/efficacy levels are expected in the intervention group compared to the control group. | 6 months
  Comparing the scale averages between groups, measuring the level of self-efficacy. Name of the Scale: Self-Efficacy Scale. Maximum 40 and minimum 8 points are taken from the scale. A high score on the scale reveals the success of not smoking even if there are encouraging factors.
The incentive factor level is expected to be lower in the intervention group than in the control group. | 6 months
  Measuring the level of incentive factor, Comparing the scale averages between groups. Name of the scale: Encouragement Factor Scale. A maximum of 40 and a minimum of 8 points can be obtained from the scale. Getting a high score from the scale; Indicates low power to stop smoking despite situations that encourage smoking
A higher level of positive health perception is expected in the intervention group than in the control group. | 6 months
  Measuring health perception, More positive health perception in the intervention group compared to the control group, unit of measure: frequency. Individuals are asked a question about how they perceive their health. Results will be compared with frequency in the intervention and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No